CLINICAL TRIAL: NCT01740999
Title: Functional Outcome in Silicone Arthroplasty Compared to Arthrodesis Screws in Patients With Osteoarthritis in the Distal Interphalangeal Joint
Brief Title: Silicone Arthroplasty vs. Arthrodesis in the Distal Interphalangeal Joint
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Non achievement of the estimated sample size of the group silicone arthroplasty in a reasonable recruitment time.
Sponsor: Schulthess Klinik (Other)
Responsible Party: Principal Investigator, Sebastian Kluge, Dr. med., Schulthess Klinik
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DIP_01
Record Dates: First submitted 2012-11-27; First posted 2012-12-04 (Estimated); Last update posted 2016-04-18 (Estimated); Status verified 2016-04

CONDITIONS: Finger Joint; Arthroplasty; Replacement
MeSH Terms: interventions — Arthrodesis

ARMS (2):
- silicone arthroplasty (Experimental): silicone arthroplasty
  Interventions: Procedure: silicone arthroplasty
- arthrodesis (Active Comparator): arthrodesis
  Interventions: Procedure: arthrodesis

INTERVENTIONS:
Procedure: silicone arthroplasty — silicone arthroplasty
  Arms: silicone arthroplasty
Procedure: arthrodesis — arthrodesis
  Arms: arthrodesis

SUMMARY:
The operational and favored standard therapy for the treatment of osteoarthritis in the distal interphalangeal joint is the arthrodesis, in which a titanium screw is used. Arthrodesis shows in the most cases the complete reduction of osteoarthritis pain and low loss of function. But restrictions are reported in fine motor skills.

The operation with silicone arthroplasty is similar. As an implant, a silicone joint is used, which has been sufficiently tested at the metacarpophalangeal joint and interphalangeal joint. The advantage of arthroplasty is the function obtained in the distal interphalangeal joint and the resulting improved fine motor skills.

ELIGIBILITY:
Inclusion Criteria:

* primary osteoarthritis in the distal interphalangeal joint
* require surgical treatment
* patient aged 18 years and over
* signed written informed consent

Exclusion Criteria:

* posttraumatic osteoarthritis
* rheumatoid disease
* pregnant woman
* any disease process that would preclude accurate evaluation (e.g. neuromuscular, psychiatric or metabolic disorder)
* legal incompetence
* no knowledge of German

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2012-06; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Michigan Hand Questionnaire (MHQ) | 12 months postoperative
  Comparison of silicone arthroplasty and arthrodesis in respect to MHQ

SECONDARY OUTCOMES:
Change of Michigan Hand Questionnaire Score | preoperative, 3mo/6mo/36mo postoperative

OTHER OUTCOMES:
Change of objective clinical parameters | preoperative, 3mo/6mo/12mo/36mo postoperative
  measurements of grip strength and range of motion

CONTACTS AND LOCATIONS:
Locations (1):
- Schulthess Klinik, Zurich, Switzerland